CLINICAL TRIAL: NCT05970341
Title: "Kidney Health: Eat Well, Live Well": A Program to Reduce Kidney Injury and Early CKD Progression Through Nutrition & Empathetic Support From a Health Partner
Brief Title: Kidney Health: Eat Well, Live Well
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Harris Health (Unknown)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, Population Health, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00002253
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: phone calls; Telehealth; Fruits and vegetables; Produce; Home delivery; grocery vouchers; gift cards; Community-based trial; Proteinuria; Diet; mental health
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Community-based randomized controlled trial stratified by self-reported diabetes diagnosis at baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research staff responsible for biomedical data collection at the sites are blinded to the participant's allocation group. Surveys are primarily self-administered on an electronic mobile device (e.g., tablet, laptop). For participants who require help reading and/or using the device, survey data will be collected via structured interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention + usual care (Experimental): 1. Welcome package
  2. Welcome information: telephone call
  3. Produce delivered at their choice of time and location + Recipes customized to produce
  4. E-gift cards to a grocery store of choice
  5. Personalized practical, emotional & educational support through a dedicated health partner
  Interventions: Behavioral: 1. Welcome package; Behavioral: 2. Welcome information (phone or text); Behavioral: 3. Produce delivery + Recipes customized to produce; Behavioral: 4. E-gift cards to a grocery store of choice; Behavioral: 5. Personalized practical & emotional support through a dedicated health partner
- Arm 2: Educational materials + usual care (Other): 1. Welcome package
  2. Welcome information: SMS/Text
  Interventions: Behavioral: 1. Welcome package; Behavioral: 2. Welcome information (phone or text)

INTERVENTIONS:
Behavioral: 1. Welcome package — At the end of the baseline data collection visit at the clinic, the Research Staff will hand the participant a welcome packet that includes:
  * educational and motivational written materials (about such topics as CKD and healthy eating for early CKD stages)
  * a collection of recipes featuring kidney-friendly vegetables
Behavioral: 2. Welcome information (phone or text) — Those allocated to the intervention arm will receive a welcome call from the Program Staff to provide further details and expectations about the program (such as delivery details and schedule).
  Those allocated to the control arm will receive an SMS text that informs them of their arm allocation, what to expect and a phone number to call for questions.
Behavioral: 3. Produce delivery + Recipes customized to produce — * Content: Bags with kidney-friendly produce will include 2 vegetables sufficient for 2 meals for 4 people, 1 type of fruit, and 1 dried fruit. The total cost is estimated at USD 20, excluding delivery, for prices in June 2022.
  * Delivery: Bags will be delivered to the participant's preferred location (e.g. home or work) and period of the day (e.g., morning, evening).
  * Recipes: SMS texts will precede each delivery to share an URL to recipes customized to the items being delivered, and to inform of an upcoming produce bag, its content.
  * Frequency:
    1. Weeks 1-2 (2 weeks): No bags delivered.
    2. Weeks 3-10 (8 weeks): Delivered weekly, for a total of 8 bags.
    3. Weeks 11-18 (8 weeks): Delivered every two weeks, for a total of 4 bags.
    4. Weeks 19-26 (8 weeks): No bags delivered.
  Arms: Arm 1: Intervention + usual care
Behavioral: 4. E-gift cards to a grocery store of choice — Five (5) e-gift cards to a major local grocery retailer chosen by the participant (from 3 options) at the following frequency:
  1. Weeks 1-6: No e-gift card.
  2. Week 7: One card of USD 30.00 value.
  3. Week 11 & 15: One card of USD 40.00, for a total of USD 80.00.
  4. Week 19 & 23: One card of USD 60.00, for a total of USD 120.00.
  Arms: Arm 1: Intervention + usual care
Behavioral: 5. Personalized practical & emotional support through a dedicated health partner — * Each participant is assigned a program staff ("dedicated health partner") who call them briefly (15 min or so) over the phone for empathy-based support on the participant's health journey, and practical suggestions for shopping and food preparation.
  * The Health Partner will share periodically via SMS text a curated list of evidence-based, trustworthy online educational resources.
  * Health partners are not trained to answer medical or health-related questions and will not provide medical guidance or advice of any kind. For such questions, they will encourage participants to contact the clinic or physician.
  * Frequency:
    1. Weeks 1-2 (2 weeks): No calls.
    2. Weeks 3-7 (4 weeks): 2 calls a week, for a total of 8 calls.
    3. Weeks 8-26 (18 weeks): 1 call every 2 weeks, for a total of 10. But during weeks 7, 11, and 19, participants will be given the choice to keep at 1x/week or decrease to 1x every 4 weeks.
  Arms: Arm 1: Intervention + usual care

SUMMARY:
This two-arm, parallel randomized trial study will assess the efficacy of a 6-month (26 weeks) community-based program in reducing kidney injury (as Urine Albumin to Creatinine ratio, uACR), cardiovascular risk (as Hemoglobin A1C and blood pressure), mental health (as PHQ-8) and diet quality (as fruits and vegetables intake and Healthy Eating Index) in community-dwelling, low-income adults diagnosed with early chronic kidney disease (stages 2 or 3 and not on kidney replacement therapies) compared to educational materials and usual care alone.

DETAILED DESCRIPTION:
This study tests a community-based program aimed at supporting adults with early-stage chronic kidney disease to change their eating habits to reduce the likelihood of kidney injury progression.

The program components were design to reduce barriers to a) eating healthier, kidney-friendly foods through the direct provision of fruits and vegetables, grocery store e-gift cards, kidney-friendly recipes, and food preparation tips; b) learning about kidney disease and the role of healthy eating in slowing its progression through educational materials; and c) social connection through empathetic relational phone calls and SMS texts from a dedicated "Health Partner".

Over a period of 6 months (26 weeks), participants randomized to the intervention arm will receive:

* kidney-friendly produce (fruits and vegetables) delivered at their preferred location
* recipes and tips on food preparation tailored to the produce
* grocery store electronic gift cards
* educational materials on CKD and disease management
* personalized practical and emotional support through a dedicated Health Partner

Researchers will see if participation in the program (intervention) reduces markers of kidney injury (Albumin:Creatinin ratio) and cardiovascular disease risk and improves diet (particularly fruits and vegetables intake) and mental health when compared to usual care (control).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Primary care visit at either one of the three partner clinics from Harris Health [Smith Clinic, Harris Health Outpatient Center (located on the LBJ campus), or Martin Luther King Jr. Health Center (MLK)] and a primary care patient within Harris Health System
* Have had at least 1 visit in the past 18 months with prior history in the clinic (i.e., not first visit)
* Diagnosis of CKD (Stage 2, 3a, and 3b) as defined by estimated Glomerular Filtration Rate (eGFR) ≥ 30 and <90 mL/min/1.73 m2 OR CDK 1 or undiagnosed with urine Albumin Creatinine Ratio ≥ 30 mg/g
* Within the past 12 months, the most current serum K+ ≤ 4.6 mEq/L
* English or Spanish speaking
* Ability to participate in the program at least 6 months
* Ability to clean, prepare, refrigerate/freeze food products that are given to them
* Have access to receive SMS text messages
* Location of preferred produce bag delivery within an available delivery zone

Exclusion Criteria:

* CKD 4, ESRD or on dialysis.
* Taking certain medications chronically (more than twice a week for 90 days) that may interfere with K+ metabolism (such as non-steroidal anti-inflammatory drugs (NSAIDs), as self-reported during enrollment screening
* Taking mineralocorticoid receptor antagonists
* Taking Warfarin
* Diagnosis of any specific kidney conditions (such as polycystic kidney disease, glomerulonephritis, Lupus associated with Nephritis, Antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV)) that would contraindicate study participation as determined by physician
* Medical history of organ transplant that would contraindicate study participation as determined by physician
* Received immunotherapy for primary or secondary kidney disease within 6 months prior to enrolment
* Diagnostic of heart failure conditions Class IV in the New York Heart Association (NYHA) functional classification
* Had myocardial infarction, unstable angina, stroke, or transient ischemic attack (TIA) within 12 weeks prior to enrolment
* Had coronary revascularization (PCI, CABG) or valvular repair within 12 weeks prior to enrolment
* On active hospice care as self-reported during enrollment screening
* Diagnosis of active malignancy requiring treatment that would contraindicate study participation as determined by physician
* Has decompensated cirrhosis as determined by physician
* Cognitive impairment that would contraindicate study participation as self-reported during enrollment screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Urine albumin:creatinine ratio (UACR) | Baseline, 3 months, 6 months
  Marker of kidney damage and a useful predictor of cardiovascular (CV) events in adults. Uses spot urine to estimate 24-hour urine albumin excretion. UACR > 30 mg/g indicates kidney damage.

SECONDARY OUTCOMES:
Hemoglobin A1C | Baseline, 3 months, 6 months
  Finger stick point-of-care portable device. Measures the average blood sugar levels over the past 3 months with a result in %. Higher A1C levels indicate poorer glycemic control and higher risk of diabetes complications.
Blood pressure (systolic/diastolic) | Baseline, 3 months, 6 months
  Direct measurement with automatic blood pressure cuff.
Food intake in the past 30 days as assessed by the Dietary Screener Questionnaire from NHANES 2009-10 | Baseline, 3 months, 6 months
  30-day food frequency questionnaire (screener) that asks for frequency of intake in the past month (per month, per week, or per day) of 28 items such as cereal, red meat, fruits and vegetables.
  This study includes four food items linked to kidney health (and mostly acid-inducing): eggs, chicken/turkey, fish, and cheese. Questions are asked in the same fashion as the other questions in the tool.
Changes in diet quality as estimates of individual mean dietary intake and frequency of fruits and vegetables consumption | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake from the Dietary Screener Questionnaire, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Reported per fruits and vegetables as cup equivalents/day.
Anxiety as measured by scores on the Generalized Anxiety Disorder 7-item (GAD-7) | Baseline, 3 months, 6 months
  Self-administered. Based on some of the DSM-V criteria for General Anxiety Disorder to identify probable cases of GAD along with measuring anxiety symptom severity. Responders are asked to rate the frequency of anxiety symptoms in the last 2 weeks on a Likert scale ranging from 0 (not at all) to 3 (nearly every day). Items are summed to provide a total score (0-21) to inform severity (1-4 minimal symptoms; 5-9 mild symptoms; 10-14 moderate symptoms; 15-21 severe symptoms).
Depressive symptoms as measured by scores on the Patient Health Questionnaire 8-item (PHQ-8) | Baseline, 3 months, 6 months
  Self-administered. Based on the nine DSM-V criteria listed under criterion A for Major Depressive Disorder. Responders are asked to rate the frequency of depression symptoms in the last 2 weeks on a Likert scale ranging from 0 (not at all) to 3 (Nearly every day). The sum of responses to each item yields a total score that screens for depression and its severity: not depressed (0-2), mild (3-5), moderate (6-8), and severe (9-12).
Loneliness measured by scores on the 3-item UCLA Loneliness Scale | Baseline, 3 months, 6 months
  Self-administered. Respondents rate each item as 'Never' , 'Rarely', 'Sometimes' or 'Often'. Scores range from 3 to 9. Higher numbers imply greater loneliness.

OTHER OUTCOMES:
Social engagement as measured by the Lubben Social Network scale 6-item | Baseline, 6 months
  Self-administered. The LSNS-6 is a self-report measure of social engagement with family and friends. The sum of the all items yields a total score that ranges between 0 and 30, with a higher score indicating more social engagement.
Perception of kidney disease and role of diet as measured by the Brief Illness Perception Questionnaire | Baseline, 6 months
  Self-administered. Answers are on a 0-10 sliding scale, except for one open-ended ranking question. Increases in item scores represent linear increases in the dimension measured.
  It contains 9 questions addressing the individual's cognitive perceptions, control over illness, beliefs about the effectiveness of treatment, experience of symptoms and emotional aspects. To better tailor it to the study population, "illness" was replaced by "kidney problem". And one question about perceived impact of food on disease was added to tailor it to the intervention.
General health and quality of life as measured by scores on the MOS Short-form 12-item (SF-12) | Baseline, 6 months
  Self-administered. Measures physical and mental health status. Summary scores range from 0-100, with higher scores indicating a better self-reported level of health.
Food security status as assessed by the USDA Food Security Survey Module: Six-Item Short Form | Baseline, 6 months
  Self-administered. Self-report assessment of access to food in the past 30 days. The sum of affirmative responses to the six questions in the module yields the household's raw score on the scale. Scores can range from 0 to 6, with higher scores indicating lower food security.
Estimated Glomerular Filtration Rate (eGFR) | As available 18 months before enrollment in the study and 15 months after study participation ends
  Obtained from Electronic Health Records. Any lab result available from 18 months prior to and 15 month post enrollment date will be obtained for study participants.
Changes in diet quality as estimates of individual mean dietary intake and frequency of dairy consumption | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Food group of dairy is reported as cup equivalents/day.
Changes in diet quality as estimates of individual mean dietary intake of added sugars | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Reported added sugars as teaspoon equivalents/day.
Changes in diet quality as estimates of individual mean dietary intake and frequency of whole grains | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Reported whole grains as ounce equivalents/day.
Changes in diet quality as estimates of individual mean dietary intake of fiber | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Reported fiber as g/day.
Changes in diet quality as estimates of individual mean dietary intake of calcium | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Reported calcium as mg/day.
Changes in diet quality as frequency of red and processed meat consumption | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. And reported red meat and processed meat as frequencies (times per day).
Changes in frequency and intake of eggs | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Added for its acid-inducing properties in chronic kidney disease. Reported as frequencies only (times per day) and amount.
Changes in frequency and intake of chicken/turkey | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Added for its acid-inducing properties in chronic kidney disease. Reported as frequencies only (times per day).
Changes in frequency and intake of fish | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Added for its association with reduced CVD risk. Reported as frequencies only (times per day).
Changes in type of cheese consumption when reported | Baseline, 3 months, 6 months
  Changes in diet quality will be measured by obtaining individual mean dietary intake, as well as frequency of food group consumption, as per analytical instructions in the National Cancer Institute, using USDA nutrient database. Soft vs. hard cheese types added for the acid-inducing properties of hard cheese in chronic kidney disease. Reported as type associated with dairy consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (3):
- United States (3):
  - Harris Health System's Outpatient Center, Houston, Texas
  - Harris Health System's Martin Luther King Jr. Health Center, Houston, Texas
  - Harris Health System's Smith Clinic, Houston, Texas

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT05970341/Prot_SAP_001.pdf